CLINICAL TRIAL: NCT02148211
Title: Fluarix/ FluLaval/ Fluarix Quadrivalent/ FluLaval Quadrivalent Pregnancy Registry: a Prospective, Exploratory, Cohort Study to Detect and Describe Abnormal Pregnancy Outcomes in Women Intentionally or Unintentionally Vaccinated With Fluarix or Fluarix Quadrivalent or FluLaval or FluLaval Quadrivalent During Pregnancy or Within 28 Days Preceding Conception.
Brief Title: Fluarix/ FluLaval/ Fluarix Quadrivalent/ FluLaval Quadrivalent Vaccine Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201476; EUPAS6521 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Results first posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Influenza
Keywords: Fluarix Quadrivalent; Fluarix; FluLaval; FluLaval Quadrivalent; Pregnancy Registry; Pregnancy outcome
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposed cohort: Pregnant women, vaccinated with any of the 4 GSK seasonal Inactivated Influenza Vaccine(s) (GSK sIIVs): Fluarix/ FluLaval/Fluarix Quadrivalent /FluLaval Quadrivalent during pregnancy or within 28 days preceding conception.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Initial and follow-up data was collected using questionnaires.

SUMMARY:
The purpose of this pregnancy registry study is to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with any of GlaxoSmithKline (GSK) Biologicals' seasonal Inactivated Influenza Vaccines (sIIVs): Fluarix, FluLaval, Fluarix Quadrivalent and FluLaval Quadrivalent.

DETAILED DESCRIPTION:
This study is a transition of existing ongoing pregnancy registries for Fluarix/ FluLaval/Fluarix Quadrivalent/ FluLaval Quadrivalent into one post-authorization safety study (PASS).

Pregnancy outcome data will be collected using questionnaires within 2 months of the estimated date of delivery (EDD) and approximately 6 months and 12 months after the EDD (for all live births) to ascertain the presence of birth defects not diagnosed before, from Q2 2014 to Q2 2019.

The intent of the Registry is to prospectively collect data such as vaccination with GSK sIIVs during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

A subject will be included in the Registry if all of the following criteria are met:

* Exposure to GSK sIIVs occurs during pregnancy or within 28 days preceding conception.
* Subject is a US resident.
* A HCP is identified (name, address and phone number).
* Subject can be identified (by GSK or HCP).

Data from registered subjects will be included in the analyses if the following criterion is met:

• Pregnancy is ongoing and the outcome is unknown at the time of initial report.

Exclusion Criteria:

Data from registered subjects will not be included in the analyses if the following criterion is met:

• Outcome of pregnancy is known at the time of initial report. Types of known outcomes include prenatal testing reports in which the results are abnormal or outside the reference range, indicating possible abnormality in the fetus.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women, residing in the US, vaccinated with any of the 4 GSK sIIVs during pregnancy or within 28 days preceding conception and who are volunteering to take part in the Pregnancy Registry before the outcome of the pregnancy is known.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Nwoji U. Seasonal influenza vaccine exposure in pregnancy: 5-year results from a pregnancy registry. Hum Vaccin Immunother. 2022 Dec 31;18(1):1932213. doi: 10.1080/21645515.2021.1932213. Epub 2021 Jun 3. PMID 34082643

RESULTS

PARTICIPANT FLOW:
Groups:
- Exposed Group: Pregnant women, vaccinated with any of the 4 GSK seasonal Inactivated Influenza Vaccine(s) (GSK sIIVs): Fluarix/ FluLaval/Fluarix Quadrivalent /FluLaval Quadrivalent during pregnancy or within 28 days preceding conception.
Period: Overall Study
Arm/Group | Exposed Group
Started | 507
Completed | 155
Not Completed | 352
Not completed — Lost to Follow-up | 352

BASELINE CHARACTERISTICS:
Groups:
- Exposure Group: Pregnant women, vaccinated with any of the 4 GSK seasonal Inactivated Influenza Vaccine(s) (GSK sIIVs): Fluarix/ FluLaval/Fluarix Quadrivalent /FluLaval Quadrivalent during pregnancy or within 28 days preceding conception.
Arm/Group | Exposure Group
Number analyzed (Participants) | 507
Age, Customized [Count of Participants; unit: Participants] — Age not specified = age unspecified in the Pregnancy Registry. Not applicable was defined as mother cases for which coding under the Pregnancy Registry was only about their infant.
  Participants
    ≤ 18 | 4
    > 18 and < 64 | 329
    Age not specified | 171
    Not applicable | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 507
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reported With Exposure and Outcomes, Stratified by Trimester of Exposure, in Pregnant Women Intentionally or Unintentionally Vaccinated With FluLaval During Pregnancy or Within 28 Days Preceding Conception
Description: Exposures and outcomes were stratified by trimester of exposure: first (1st), second (2nd), third (3rd) and unknown trimester (Tr?) multiple exposures during a pregnancy were classified by the earliest trimester of exposure. The estimated gestational age at the time of vaccination was calculated based on the date of the last menstrual period. The 2nd trimester was considered to begin at week 14 and the 3rd trimester begun at week 28. The presence or absence of birth defects or other abnormalities was evaluated within each of the preceding outcome categories. Ongoing = subject still pregnant at the time of last contact. Note: The remaining pregnancies were ongoing at the time of last contact by the study staff. No further information on the outcome of these pregnancies was available as of 1st April 2020. Unknown = unknown outcome at the time of last contact.
Time Frame: Data collected for a minimum of 5 years starting from June 1, 2014 till May 31, 2019: for each subject, data was collected within 2 months of estimated date of delivery (EDD) and follow-up 6 and 12 months after EDD (for all live births)
Population: Analysis was performed on pregnant women vaccinated with FluLaval vaccine during pregnancy or within 28 days preceding conception who volunteered to take part of the study and who completed the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 8
Participants
  Ongoing, 1st Tr. | 2
  Ongoing, 2nd Tr. | 3
  Ongoing, 3rd Tr. | 0
  Ongoing, Tr? | 1
  Unknown, 1st Tr. | 0
  Unknown, 2nd Tr. | 0
  Unknown, 3rd Tr. | 2
  Unknown, Tr? | 0

2. Primary Outcome: Number of Subjects Reported With Exposure and Outcomes, Stratified by Trimester of Exposure in Pregnant Women Intentionally or Unintentionally Vaccinated With FluLaval Quadrivalent During Pregnancy or Within 28 Days Preceding Conception
Description: Exposure and outcomes were stratified by trimester of exposure: 1st, 2nd, 3rd and Tr?; multiple exposures during a pregnancy were classified by the earliest trimester of exposure. The estimated gestational age at the time of vaccination was calculated as described in the first outcome. Results were presented for the following categories: Ongoing, Live infants without congenital anomalies (Live infants without CA.); Spontaneous abortions with no apparent congenital anomalies (Sp. abortions with no ACA); Spontaneous abortions with congenital anomalies (Sp. abortions with CA). One subject had FluLaval Quadrivalent and Fluarix Quadrivalent listed as vaccine used. Therefore, same case was included in the respective table of each product in "Live infants without CA, 3rd Tr." category. Note: The remaining pregnancies were ongoing at the time of last contact by the study staff. No further information on the outcome of these pregnancies was available as of 1st April 2020.
Time Frame: as for outcome 1
Population: Analysis was performed on pregnant women vaccinated with FluLaval Quadrivalent vaccine during pregnancy or within 28 days preceding conception who volunteered to take part of the study, and who completed the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 33
Participants
  Ongoing, 1st Tr. | 0
  Ongoing, 2nd Tr. | 1
  Ongoing, 3rd Tr. | 1
  Ongoing, Tr? | 6
  Live infants without CA, 1st Tr. | 4
  Live infants without CA, 2nd Tr. | 6
  Live infants without CA, 3rd Tr. | 10
  Live infants without CA, Tr? | 3
  Sp. abortions with no ACA, 1st Tr. | 0
  Sp. abortions with no ACA, 2nd Tr. | 0
  Sp. abortions with no ACA, 3rd Tr. | 0
  Sp. abortions with no ACA, Tr? | 1
  Sp. abortions with CA, 1st Tr. | 1
  Sp. abortions with CA, 2nd Tr. | 0
  Sp. abortions with CA, 3rd Tr. | 0
  Sp. abortions with CA, Tr? | 0

3. Primary Outcome: Number of Subjects Reported With Exposure and Outcomes, Stratified by Trimester of Exposure in Pregnant Women Intentionally or Unintentionally Vaccinated With Fluarix During Pregnancy or Within 28 Days Preceding Conception
Description: Exposure and outcomes were stratified by trimester of exposure: 1st, 2nd, 3rd and Tr?; multiple exposures during a pregnancy were classified by the earliest trimester of exposure. The estimated gestational age at the time of vaccination was calculated as described in the first outcome. Unknown = unknown outcome at the time of last contact.
Time Frame: as for outcome 1
Population: Analysis was performed on pregnant women vaccinated with Fluarix vaccine during pregnancy or within 28 days preceding conception who volunteered to take part of the study, and who completed the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 1
Participants
  Unknown, 1st Tr. | 0
  Unknown, 2nd Tr. | 0
  Unknown, 3rd Tr. | 0
  Unknown, Tr? | 1

4. Primary Outcome: Number of Subjects Reported With Exposure and Outcomes Stratified by Trimester of Exposure in Pregnant Women Intentionally or Unintentionally Vaccinated With Fluarix Quadrivalent During Pregnancy or Within 28 Days Preceding Conception
Description: Exposure and outcomes were stratified by trimester of exposure: 1st, 2nd, 3rd and Tr?; multiple exposures during a pregnancy were classified by the earliest trimester of exposure. The estimated gestational age at the time of vaccination was calculated as described in the first outcome. Results were presented for the following categories: Ongoing, Live infants without CA; Live infants with CA; Sp. abortions with no ACA; Sp. abortions with CA; Stillbirth with no ACA. Unknown = unknown pregnancy outcome at the time of last contact. One subject had FluLaval Quadrivalent and Fluarix Quadrivalent listed as vaccine used. Therefore, same case was included in the respective table of each product in "Live infants without CA, 3rd Tr." category. Note: The remaining pregnancies were ongoing at the time of last contact by the study staff. No further information on the outcome of these pregnancies was available as of 1st April 2020.
Time Frame: as for outcome 1
Population: Analysis was performed on pregnant women vaccinated with Fluarix Quadrivalent vaccine during pregnancy or within 28 days preceding conception who volunteered to take part of the study, and who completed the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 114
Participants
  Ongoing, 1st Tr. | 5
  Ongoing, 2nd Tr. | 2
  Ongoing, 3rd Tr. | 4
  Ongoing, Tr? | 15
  Live infants without CA, 1st Tr. | 15
  Live infants without CA, 2nd Tr. | 31
  Live infants without CA, 3rd Tr. | 21
  Live infants without CA, Tr? | 12
  Live infants with CA, 1st Tr. | 0
  Live infants with CA, 2nd Tr. | 3
  Live infants with CA, 3rd Tr. | 0
  Live infants with CA, Tr? | 0
  Sp. abortions with no ACA, 1st Tr. | 1
  Sp. abortions with no ACA, 2nd Tr. | 0
  Sp. abortions with no ACA, 3rd Tr. | 0
  Sp. abortions with no ACA, Tr? | 0
  Sp. abortions with CA, 1st Tr. | 0
  Sp. abortions with CA, 2nd Tr. | 0
  Sp. abortions with CA, 3rd Tr. | 0
  Sp. abortions with CA, Tr? | 0
  Stillbirth with no ACA, 1st Tr. | 1
  Stillbirth with no ACA, 2nd Tr. | 0
  Stillbirth with no ACA, 3rd Tr. | 0
  Stillbirth with no ACA, Tr? | 0
  Unknown, 1st Tr. | 1
  Unknown, 2nd Tr. | 0
  Unknown, 3rd Tr. | 0
  Unknown, Tr? | 3

5. Primary Outcome: Number of Subjects Reported With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product during the clinical study. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Data collected for a minimum of 5 years starting from June 1, 2014 till May 31, 2019
Population: Analysis was performed on pregnant women vaccinated with GSK sIIV vaccine during pregnancy or within 28 days preceding conception who volunteered to take part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 507
Participants | 507

6. Primary Outcome: Number of Subjects Reported With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Data collected for a minimum of 5 years starting from June 1, 2014 till May 31, 2019
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 507
Participants | 9

ADVERSE EVENTS:
Time Frame: Data collected for a minimum of 5 years starting from June 1, 2014 till May 31, 2019
Description: All-cause mortality reported data are fetal deaths. Only unanticipated AEs were collected in the study. Anticipated AEs were not assessed/monitored.
Arm/Group | Exposure Group
All-Cause Mortality (participants affected / at risk) | 2/507
Serious Adverse Events (participants affected / at risk) | 9/507
Other Adverse Events (participants affected / at risk) | 507/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exposure Group (N=507)
Cleft lip and palate (Congenital, familial and genetic disorders) | 1 (1) — This SAE is reported in infant.
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 (1) — This SAE is reported in infant.
Injection site cellulitis (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exposure Group (N=507)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Crying (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site edema (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Injection site warmth (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Multiple allergies (Immune system disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Contraindicated product administered (Injury, poisoning and procedural complications) | 1 (1)
Expired product administered (Injury, poisoning and procedural complications) | 5 (5)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 503 (504) — The inclusion of this in the AE table is a function of the coding convention of the medical coding system.
Exposure via body fluid (Injury, poisoning and procedural complications) | 1 (1)
Extra dose administered (Injury, poisoning and procedural complications) | 10 (10)
Maternal exposure before pregnancy (Injury, poisoning and procedural complications) | 1 (1) — The inclusion of this in the AE table is a function of the coding convention of the medical coding system.
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 2 (2) — The inclusion of this in the AE table is a function of the coding convention of the medical coding system.
Maternal exposure timing unspecified (Injury, poisoning and procedural complications) | 1 (1) — The inclusion of this in the AE table is a function of the coding convention of the medical coding system.
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Wrong product administered (Injury, poisoning and procedural complications) | 5 (5)
Wrong technique in product usage process (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Arrested labor (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Live birth (Pregnancy, puerperium and perinatal conditions) | 103 (103)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 4 (4)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT02148211/Prot_SAP_000.pdf